CLINICAL TRIAL: NCT06536413
Title: Phase IB/II Study Combining All-Trans Retinoic Acid (ATRA) With Carfilzomib Based Therapy in Plasma Cell Myeloma Patients Refractory to Carfilzomib
Brief Title: ATRA and Carfilzomib in Plasma Cell Myeloma Patients
Acronym: ATRA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Sai Ravi Kiran Pingali, Hematologist-Oncologist, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00037762 (HMCC-HM22-001)
Record Dates: First submitted 2024-06-27; First posted 2024-08-05 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All-Trans Retinoic Acid (ATRA), Carfilzomib, and Dexamethasone (Experimental): Carfilzomib will be given at Cycle 1 (20 mg/m2 on Days 1, 70 mg/m2 on Days 8 and 15) and Cycles 2 - onward (70 mg/m2 on Days 1, 8, and 15) as a 30-minute intravenous (IV) infusion to evaluate tolerability to treatment.
  Dexamethasone will be given [20 mg, PO/IV] on the days of carfilzomib treatment.
  ATRA will be given for 3 weeks (21 days) out of every 4 weeks (28 days) up to a maximum of 24 weeks (6 cycles). Only for Cycle 1, patients will start oral ATRA 25 mg/m2 7 days prior to Cycle 1 Day 1 through Cycle 1 Day 21 for a total of 28 days of dosing.
  To assign a dose to the next cohort of patients, dose escalation/de-escalation according to the trials Bayesian Optimal Interval (BOIN) Design is conducted. In patients who respond and do not have any dose limiting toxicity (DLT), treatment will continue for a total of 6 cycles in the phase II expansion cohort and subsequently transitioned to standard -of-care options.
  Interventions: Drug: All-Trans Retinoic Acid (ATRA) Dose 0; Drug: All-Trans Retinoic Acid (ATRA) Dose -1; Drug: All-Trans Retinoic Acid (ATRA) Dose 1

INTERVENTIONS:
Drug: All-Trans Retinoic Acid (ATRA) Dose 0 — Patients will receive oral ATRA 25 mg/m2 per day in two divided doses with carfilzomib-based regimens.
  Eligible patients will enter the study in cohorts of two with the first cohort treated at Dose 0. To assign a dose to the next cohort of patients, dose escalation/de-escalation according to the the trials Bayesian Optimal Interval (BOIN) Design is conducted. In patients who respond and do not have any dose limiting toxicity (DLT), treatment will continue for a total of 6 cycles in the phase II expansion cohort and subsequently transitioned to standard -of-care options. Each cycle will be 28 days. In phase 1b, a minimum of 16 evaluable patients will be recruited and in the second phase a minimum of 26 evaluable patients will be recruited. A minimum of 42 evaluable patients will be recruited in the study.
  If a dose limiting toxicity occurs at 25 mg/m2, then the dose will be reduced by 50% to 15 mg/sq m daily in two divided doses.
Drug: All-Trans Retinoic Acid (ATRA) Dose -1 — Patients will receive oral ATRA 15 mg/m2 per day in two divided doses with carfilzomib-based regimens.
  Eligible patients will enter the study in cohorts of two with the first cohort treated at Dose 0. To assign a dose to the next cohort of patients, dose escalation/de-escalation according to the trials Bayesian Optimal Interval (BOIN) Design is conducted. In patients who respond and do not have any dose limiting toxicity (DLT), treatment will continue for a total of 6 cycles in the phase II expansion cohort and subsequently transitioned to standard -of-care options. Each cycle will be 28 days. In phase 1b, a minimum of 16 evaluable patients will be recruited and in the second phase a minimum of 26 evaluable patients will be recruited. A minimum of 42 evaluable patients will be recruited in the study.
Drug: All-Trans Retinoic Acid (ATRA) Dose 1 — Patients will receive oral ATRA 45 mg/m2 per day in two divided doses with carfilzomib-based regimens.
  Eligible patients will enter the study in cohorts of two with the first cohort treated at Dose 0. To assign a dose to the next cohort of patients, dose escalation/de-escalation according to the trials Bayesian Optimal Interval (BOIN) Design is conducted. In patients who respond and do not have any dose limiting toxicity (DLT), treatment will continue for a total of 6 cycles in the phase II expansion cohort and subsequently transitioned to standard -of-care options. Each cycle will be 28 days. In phase 1b, a minimum of 16 evaluable patients will be recruited and in the second phase a minimum of 26 evaluable patients will be recruited. A minimum of 42 evaluable patients will be recruited in the study.

SUMMARY:
This is a Phase IB/II trial that will investigate the safety, tolerability and efficacy of combination therapy using All-Trans Retinoic Acid (ATRA) with Carfilzomib based therapies in plasma cell myeloma also commonly referred as Multiple Myeloma (MM), in patients considered refractory to proteasome inhibitors (PIs). Multiple myeloma is an incurable clonal plasma cell disorder that comprises 10% of all hematologic malignancies. Over the past 30 years the global prevalence of multiple myeloma has risen to 126%, with 85% of diagnoses occurring in patients >55 years of age. In the past 15 years, survival has improved considerably, which is attributed to the development of multiple different classes of medications, including proteasome inhibitors. Proteasome inhibitors are the foundation of many multiple myeloma treatments in both transplant eligible and ineligible patients for the past 2 decades. While proteasome inhibitors have improved both progression free survival (PFS) and overall survival (OS), many patients eventually develop disease progression arising from resistance to therapies. As a result, there is an unmet need to overcome resistance and find ways to enhance multiple myeloma sensitivity to proteasome inhibitor toxicity. Carfilzomib, a modified peptide epoxyketone that selectively targets intracellular proteasome enzymes, is approved in combination with dexamethasone in patients that have received ≥1 line of therapy or in combination. There are few studies assessing ways to enhance carfilzomib-mediated multiple myeloma toxicity. All-Trans Retinoic Acid (ATRA) is an oxidative metabolite of retinol (vitamin A) and plays an important role in the regulation of cellular proliferation and differentiation. In a recent pre-clinical study, ATRA was found to enhance sensitivity of carfilzomib-mediated apoptosis in vitro via an interferon beta (IFN-β) response pathway. In the clinical setting, ATRA is a well-tolerated drug that has shown little change in the rate of adverse events in early clinical trials with multiple myeloma. The investigators hypothesize that ATRA enhances sensitivity of multiple myeloma to carfilzomib therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years with relapsed/refractory multiple myeloma documented according to International Myeloma Working Group (IMWG) criteria.
2. Previously treated with at least three lines of therapy which would include Immunomodulatory drugs (IMiDs), Proteosome inhibitors (including carfilzomib), anti-CD 38 antibodies and failed to achieve a minor response after completing at least 2 cycles of carfilzomib-based therapy or are relapsed while on therapy.
3. Patient or legal guardian voluntarily can sign informed consent.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 2
5. Adequate organ function defined as:

   1. Hemoglobin ≥8 g/dL (baseline or after Peripheral Red Blood Cell transfusion), Platelet count >75,000 and Absolute Neutrophil Count >1000/ micro liter.
   2. Left Ventricular Ejection fraction ≥50%
   3. Creatinine Clearance ≥ 30 ml/min
   4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN)
   5. Total bilirubin ≤ 1.5 × ULN
6. Measurable disease requiring treatment defined as patients having one or more of the criteria below:

   1. Serum M protein ≥ 0.5 g/dL or
   2. Urine M-protein ≥ 200 mg/24 hours or
   3. Serum free light chain (SFLC) ≥ 100 mg/L (involved light chain) and an abnormal serum
   4. kappa lambda ratio.
7. If previous autologous stem cell transplantation, must have fully recovered from transplant related toxicities and be >60 days from transplant and have had hematologic recovery independent of growth factor support.
8. Willingness to undergo interim bone marrow biopsy as scheduled or if felt to be medically indicated.
9. Life Expectancy ≥ 6 months
10. Women with childbearing potential and men should practice at least one of the following methods of birth control:

    1. Total abstinence from sexual intercourse (periodic abstinence not acceptable);
    2. Surgically sterile partner(s) including vasectomy, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy;
    3. Intrauterine device with an additional method of contraception to make two effective methods of contraception during treatment with Vesanoid;
    4. Double-barrier method (condom + diaphragm or cervical cap with spermicide, contraceptive sponge, jellies, or cream);
    5. Hormonal contraceptives (oral, parenteral, vaginal ring, or transdermal) for at least 3 months prior to study drug administration. If hormonal contraceptives are used, the specific contraceptive must have been used for at least 3 months prior to study drug administration. If the patient is currently using a hormonal contraceptive, she should also use a barrier method during this study Women of child-bearing potential must have a negative results of a pregnancy test performed at initial screening on a serum sample obtained within 21 days prior to C1D1, and prior to dosing on a urine sample obtained within 72 hours of the first study drug administration. Males must refrain from sperm donations from date of C1D1 to 90 days after the last date of the study drug.

Exclusion Criteria:

1. Non-secretory or hyposecretory multiple myeloma, defined as <0.5 g/dL M-protein in serum, <200 mg/24-hour urine M-protein, or disease only measured by serum free light chain.
2. Plasma Cell Leukemia (Previously treated Plasma Cell Leukemia can be included per PI discretion)
3. Concurrent light chain amyloidosis
4. Central nervous system involvement (patients with known brain metastases have poor prognosis and often develop progressive neurologic dysfunction that may confound the evaluation of neurologic and other Adverse Events while on ATRA).
5. Pregnant or breast feeding
6. Severe, active, recurrent, or intercurrent infection (viral, bacterial, fungal), or diagnosis of neutropenia and fever within one week of C1D1.
7. History of Allogeneic hematopoietic cell transplantation or solid organ transplantation.
8. Unstable angina pectoris, cardiac arrhythmia or > New York Heart Failure association class II cardiac failure, defined as comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or anginal pain.
9. Patient has a significant history of renal, neurologic (peripheral neuropathy), psychiatric, endocrinologic (diabetes mellitus), metabolic, immunologic, cardiovascular, pulmonary, hepatic disease, or significant social situation within the past 6 months that, in the opinion of the investigator, would impede his/her ability to fully participate in the study. For patients who have required an intervention for the above diseases within the past 6 months, a case-by-case discussion with the investigator must occur.
10. On investigational therapies within 12 weeks of enrollment.
11. Previous allergic reaction or intolerance to a proteasome inhibitor, including carfilzomib, bortezomib, or ixazomib.
12. Or deemed unfit for the study on evaluation by Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of ATRA in combination with Carfilzomib/ Dexamethazone and RP2D | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws from the study, whichever came first, assessed up to 7 months.
  To determine safety and tolerability of ATRA in combination with carfilzomib/dexamethasone and determine the recommended phase II dose (RP2D). The RP2D will be defined as the highest dose administered at which 6 patients are treated with with no more than 2 experiencing dose limiting toxicity (DLT) (determined by diseases progression, unacceptable toxicity, physician's discretion).

SECONDARY OUTCOMES:
Efficacy of combination therapy of ATRA, Carfilzomib, and Dexamethasone in resistant Multiple Myeloma | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws, whichever came first, assessed up to 7 months.
  Overall Response Rate (percentage of patients with complete response [CR] or partial response [PR]), as defined by International Myeloma Working Group (IMWG) criteria.
Duration of Response of combination therapy of ATRA, Carfilzomib, and Dexamethasone in resistant Multiple Myeloma | From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease, whichever came first, assessed up to 7 months after initial treatment date.
  Duration of response rate as defined by the duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | The dose limiting toxicity period begins from date of initial treatment until 21 days after.
  Toxicity and safety, as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Disease response as measured by serum, viable cryopreserved peripheral blood mononuclear cells, and bone marrow myeloma plasma cells. | Correlative samples will be collected at Baseline, Cycle 1 Day 1, Cycle 2 Day 1, and Cycle 3 Day 1. Cycles are 28 days in length.
  To characterize the disease response of the ATRA and carfilzomib/dexamethasone combination as measured by serum, viable cryopreserved peripheral blood mononuclear cells, and bone marrow myeloma plasma cells.

CONTACTS AND LOCATIONS:
Overall Officials: Sai Ravi Pingali, MD, Principal Investigator — Houston Methodist Neal Cancer Center
Locations (1):
- Houston Methodist Neal Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Otsuki T, Sakaguchi H, Hatayama T, Wu P, Takata A, Hyodoh F. Effects of all-trans retinoic acid (ATRA) on human myeloma cells. Leuk Lymphoma. 2003 Oct;44(10):1651-6. doi: 10.1080/1042819031000099652. PMID 14692515
- [Background] Nijhof IS, Groen RW, Lokhorst HM, van Kessel B, Bloem AC, van Velzen J, de Jong-Korlaar R, Yuan H, Noort WA, Klein SK, Martens AC, Doshi P, Sasser K, Mutis T, van de Donk NW. Upregulation of CD38 expression on multiple myeloma cells by all-trans retinoic acid improves the efficacy of daratumumab. Leukemia. 2015 Oct;29(10):2039-49. doi: 10.1038/leu.2015.123. Epub 2015 May 15. PMID 25975191
- [Background] Frerichs KA, Minnema MC, Levin MD, Broijl A, Bos GMJ, Kersten MJ, Mutis T, Verkleij CPM, Nijhof IS, Maas-Bosman PWC, Klein SK, Zweegman S, Sonneveld P, van de Donk NWCJ. Efficacy and safety of daratumumab combined with all-trans retinoic acid in relapsed/refractory multiple myeloma. Blood Adv. 2021 Dec 14;5(23):5128-5139. doi: 10.1182/bloodadvances.2021005220. PMID 34625791
- [Background] Garcia-Guerrero E, Rodriguez-Lobato LG, Sierro-Martinez B, Danhof S, Bates S, Frenz S, Haertle L, Gotz R, Sauer M, Rasche L, Kortum KM, Perez-Simon JA, Einsele H, Hudecek M, Prommersberger SR. All-trans retinoic acid works synergistically with the gamma-secretase inhibitor crenigacestat to augment BCMA on multiple myeloma and the efficacy of BCMA-CAR T cells. Haematologica. 2023 Feb 1;108(2):568-580. doi: 10.3324/haematol.2022.281339. PMID 36722406
- [Background] Wang Q, Lin Z, Wang Z, Ye L, Xian M, Xiao L, Su P, Bi E, Huang YH, Qian J, Liu L, Ma X, Yang M, Xiong W, Zu Y, Pingali SR, Xu B, Yi Q. RARgamma activation sensitizes human myeloma cells to carfilzomib treatment through the OAS-RNase L innate immune pathway. Blood. 2022 Jan 6;139(1):59-72. doi: 10.1182/blood.2020009856. PMID 34411225
- [Background] Landgren O, Kyle RA, Pfeiffer RM, Katzmann JA, Caporaso NE, Hayes RB, Dispenzieri A, Kumar S, Clark RJ, Baris D, Hoover R, Rajkumar SV. Monoclonal gammopathy of undetermined significance (MGUS) consistently precedes multiple myeloma: a prospective study. Blood. 2009 May 28;113(22):5412-7. doi: 10.1182/blood-2008-12-194241. Epub 2009 Jan 29. PMID 19179464
- [Background] Kyle RA, Therneau TM, Rajkumar SV, Larson DR, Plevak MF, Offord JR, Dispenzieri A, Katzmann JA, Melton LJ 3rd. Prevalence of monoclonal gammopathy of undetermined significance. N Engl J Med. 2006 Mar 30;354(13):1362-9. doi: 10.1056/NEJMoa054494. PMID 16571879
- [Background] Rajkumar SV, Dimopoulos MA, Palumbo A, Blade J, Merlini G, Mateos MV, Kumar S, Hillengass J, Kastritis E, Richardson P, Landgren O, Paiva B, Dispenzieri A, Weiss B, LeLeu X, Zweegman S, Lonial S, Rosinol L, Zamagni E, Jagannath S, Sezer O, Kristinsson SY, Caers J, Usmani SZ, Lahuerta JJ, Johnsen HE, Beksac M, Cavo M, Goldschmidt H, Terpos E, Kyle RA, Anderson KC, Durie BG, Miguel JF. International Myeloma Working Group updated criteria for the diagnosis of multiple myeloma. Lancet Oncol. 2014 Nov;15(12):e538-48. doi: 10.1016/S1470-2045(14)70442-5. Epub 2014 Oct 26. PMID 25439696
- [Background] Kyle RA, Remstein ED, Therneau TM, Dispenzieri A, Kurtin PJ, Hodnefield JM, Larson DR, Plevak MF, Jelinek DF, Fonseca R, Melton LJ 3rd, Rajkumar SV. Clinical course and prognosis of smoldering (asymptomatic) multiple myeloma. N Engl J Med. 2007 Jun 21;356(25):2582-90. doi: 10.1056/NEJMoa070389. PMID 17582068
- [Background] Cowan AJ, Allen C, Barac A, Basaleem H, Bensenor I, Curado MP, Foreman K, Gupta R, Harvey J, Hosgood HD, Jakovljevic M, Khader Y, Linn S, Lad D, Mantovani L, Nong VM, Mokdad A, Naghavi M, Postma M, Roshandel G, Shackelford K, Sisay M, Nguyen CT, Tran TT, Xuan BT, Ukwaja KN, Vollset SE, Weiderpass E, Libby EN, Fitzmaurice C. Global Burden of Multiple Myeloma: A Systematic Analysis for the Global Burden of Disease Study 2016. JAMA Oncol. 2018 Sep 1;4(9):1221-1227. doi: 10.1001/jamaoncol.2018.2128. PMID 29800065
- [Background] Minnie SA, Hill GR. Immunotherapy of multiple myeloma. J Clin Invest. 2020 Apr 1;130(4):1565-1575. doi: 10.1172/JCI129205. PMID 32149732
- [Background] Ito S. Proteasome Inhibitors for the Treatment of Multiple Myeloma. Cancers (Basel). 2020 Jan 22;12(2):265. doi: 10.3390/cancers12020265. PMID 31979059
- [Background] Herndon TM, Deisseroth A, Kaminskas E, Kane RC, Koti KM, Rothmann MD, Habtemariam B, Bullock J, Bray JD, Hawes J, Palmby TR, Jee J, Adams W, Mahayni H, Brown J, Dorantes A, Sridhara R, Farrell AT, Pazdur R. U.s. Food and Drug Administration approval: carfilzomib for the treatment of multiple myeloma. Clin Cancer Res. 2013 Sep 1;19(17):4559-63. doi: 10.1158/1078-0432.CCR-13-0755. Epub 2013 Jun 17. PMID 23775332
- [Background] Stewart AK, Rajkumar SV, Dimopoulos MA, Masszi T, Spicka I, Oriol A, Hajek R, Rosinol L, Siegel DS, Mihaylov GG, Goranova-Marinova V, Rajnics P, Suvorov A, Niesvizky R, Jakubowiak AJ, San-Miguel JF, Ludwig H, Wang M, Maisnar V, Minarik J, Bensinger WI, Mateos MV, Ben-Yehuda D, Kukreti V, Zojwalla N, Tonda ME, Yang X, Xing B, Moreau P, Palumbo A; ASPIRE Investigators. Carfilzomib, lenalidomide, and dexamethasone for relapsed multiple myeloma. N Engl J Med. 2015 Jan 8;372(2):142-52. doi: 10.1056/NEJMoa1411321. Epub 2014 Dec 6. PMID 25482145
- [Background] Dimopoulos MA, Moreau P, Palumbo A, Joshua D, Pour L, Hajek R, Facon T, Ludwig H, Oriol A, Goldschmidt H, Rosinol L, Straub J, Suvorov A, Araujo C, Rimashevskaya E, Pika T, Gaidano G, Weisel K, Goranova-Marinova V, Schwarer A, Minuk L, Masszi T, Karamanesht I, Offidani M, Hungria V, Spencer A, Orlowski RZ, Gillenwater HH, Mohamed N, Feng S, Chng WJ; ENDEAVOR Investigators. Carfilzomib and dexamethasone versus bortezomib and dexamethasone for patients with relapsed or refractory multiple myeloma (ENDEAVOR): a randomised, phase 3, open-label, multicentre study. Lancet Oncol. 2016 Jan;17(1):27-38. doi: 10.1016/S1470-2045(15)00464-7. Epub 2015 Dec 5. PMID 26671818
- [Background] Moreau P, Mateos MV, Berenson JR, Weisel K, Lazzaro A, Song K, Dimopoulos MA, Huang M, Zahlten-Kumeli A, Stewart AK. Once weekly versus twice weekly carfilzomib dosing in patients with relapsed and refractory multiple myeloma (A.R.R.O.W.): interim analysis results of a randomised, phase 3 study. Lancet Oncol. 2018 Jul;19(7):953-964. doi: 10.1016/S1470-2045(18)30354-1. Epub 2018 Jun 1. PMID 29866475
- [Background] Obeng EA, Carlson LM, Gutman DM, Harrington WJ Jr, Lee KP, Boise LH. Proteasome inhibitors induce a terminal unfolded protein response in multiple myeloma cells. Blood. 2006 Jun 15;107(12):4907-16. doi: 10.1182/blood-2005-08-3531. Epub 2006 Feb 28. PMID 16507771
- [Background] Mitsiades N, Mitsiades CS, Poulaki V, Chauhan D, Fanourakis G, Gu X, Bailey C, Joseph M, Libermann TA, Treon SP, Munshi NC, Richardson PG, Hideshima T, Anderson KC. Molecular sequelae of proteasome inhibition in human multiple myeloma cells. Proc Natl Acad Sci U S A. 2002 Oct 29;99(22):14374-9. doi: 10.1073/pnas.202445099. Epub 2002 Oct 21. PMID 12391322
- [Background] Yarde DN, Oliveira V, Mathews L, Wang X, Villagra A, Boulware D, Shain KH, Hazlehurst LA, Alsina M, Chen DT, Beg AA, Dalton WS. Targeting the Fanconi anemia/BRCA pathway circumvents drug resistance in multiple myeloma. Cancer Res. 2009 Dec 15;69(24):9367-75. doi: 10.1158/0008-5472.CAN-09-2616. PMID 19934314
- [Background] Robak P, Drozdz I, Szemraj J, Robak T. Drug resistance in multiple myeloma. Cancer Treat Rev. 2018 Nov;70:199-208. doi: 10.1016/j.ctrv.2018.09.001. Epub 2018 Sep 4. PMID 30245231
- [Background] Verbrugge SE, Assaraf YG, Dijkmans BA, Scheffer GL, Al M, den Uyl D, Oerlemans R, Chan ET, Kirk CJ, Peters GJ, van der Heijden JW, de Gruijl TD, Scheper RJ, Jansen G. Inactivating PSMB5 mutations and P-glycoprotein (multidrug resistance-associated protein/ATP-binding cassette B1) mediate resistance to proteasome inhibitors: ex vivo efficacy of (immuno)proteasome inhibitors in mononuclear blood cells from patients with rheumatoid arthritis. J Pharmacol Exp Ther. 2012 Apr;341(1):174-82. doi: 10.1124/jpet.111.187542. Epub 2012 Jan 10. PMID 22235146
- [Background] Chen X, Rotenberg SA. PhosphoMARCKS drives motility of mouse melanoma cells. Cell Signal. 2010 Jul;22(7):1097-103. doi: 10.1016/j.cellsig.2010.03.003. Epub 2010 Mar 6. PMID 20211725
- [Background] Finlayson AE, Freeman KW. A cell motility screen reveals role for MARCKS-related protein in adherens junction formation and tumorigenesis. PLoS One. 2009 Nov 18;4(11):e7833. doi: 10.1371/journal.pone.0007833. PMID 19924305
- [Background] Li T, Li D, Sha J, Sun P, Huang Y. MicroRNA-21 directly targets MARCKS and promotes apoptosis resistance and invasion in prostate cancer cells. Biochem Biophys Res Commun. 2009 Jun 5;383(3):280-5. doi: 10.1016/j.bbrc.2009.03.077. Epub 2009 Mar 18. PMID 19302977
- [Background] Micallef J, Taccone M, Mukherjee J, Croul S, Busby J, Moran MF, Guha A. Epidermal growth factor receptor variant III-induced glioma invasion is mediated through myristoylated alanine-rich protein kinase C substrate overexpression. Cancer Res. 2009 Oct 1;69(19):7548-56. doi: 10.1158/0008-5472.CAN-08-4783. Epub 2009 Sep 22. PMID 19773446
- [Background] Franke NE, Kaspers GL, Assaraf YG, van Meerloo J, Niewerth D, Kessler FL, Poddighe PJ, Kole J, Smeets SJ, Ylstra B, Bi C, Chng WJ, Horton TM, Menezes RX, Musters RJ, Zweegman S, Jansen G, Cloos J. Exocytosis of polyubiquitinated proteins in bortezomib-resistant leukemia cells: a role for MARCKS in acquired resistance to proteasome inhibitors. Oncotarget. 2016 Nov 15;7(46):74779-74796. doi: 10.18632/oncotarget.11340. PMID 27542283
- [Background] Morito N, Yoh K, Maeda A, Nakano T, Fujita A, Kusakabe M, Hamada M, Kudo T, Yamagata K, Takahashi S. A novel transgenic mouse model of the human multiple myeloma chromosomal translocation t(14;16)(q32;q23). Cancer Res. 2011 Jan 15;71(2):339-48. doi: 10.1158/0008-5472.CAN-10-1057. Epub 2011 Jan 11. PMID 21224354
- [Background] Besse A, Stolze SC, Rasche L, Weinhold N, Morgan GJ, Kraus M, Bader J, Overkleeft HS, Besse L, Driessen C. Carfilzomib resistance due to ABCB1/MDR1 overexpression is overcome by nelfinavir and lopinavir in multiple myeloma. Leukemia. 2018 Feb;32(2):391-401. doi: 10.1038/leu.2017.212. Epub 2017 Jul 5. PMID 28676669
- [Background] Zheng Z, Liu T, Zheng J, Hu J. Clarifying the molecular mechanism associated with carfilzomib resistance in human multiple myeloma using microarray gene expression profile and genetic interaction network. Onco Targets Ther. 2017 Mar 1;10:1327-1334. doi: 10.2147/OTT.S130742. eCollection 2017. PMID 28280367
- [Background] Baranowska K, Misund K, Starheim KK, Holien T, Johansson I, Darvekar S, Buene G, Waage A, Bjorkoy G, Sundan A. Hydroxychloroquine potentiates carfilzomib toxicity towards myeloma cells. Oncotarget. 2016 Oct 25;7(43):70845-70856. doi: 10.18632/oncotarget.12226. PMID 27683126
- [Background] Waldschmidt JM, Simon A, Wider D, Muller SJ, Follo M, Ihorst G, Decker S, Lorenz J, Chatterjee M, Azab AK, Duyster J, Wasch R, Engelhardt M. CXCL12 and CXCR7 are relevant targets to reverse cell adhesion-mediated drug resistance in multiple myeloma. Br J Haematol. 2017 Oct;179(1):36-49. doi: 10.1111/bjh.14807. Epub 2017 Jul 2. PMID 28670693
- [Background] Vogl DT, Stadtmauer EA, Tan KS, Heitjan DF, Davis LE, Pontiggia L, Rangwala R, Piao S, Chang YC, Scott EC, Paul TM, Nichols CW, Porter DL, Kaplan J, Mallon G, Bradner JE, Amaravadi RK. Combined autophagy and proteasome inhibition: a phase 1 trial of hydroxychloroquine and bortezomib in patients with relapsed/refractory myeloma. Autophagy. 2014 Aug;10(8):1380-90. doi: 10.4161/auto.29264. Epub 2014 May 20. PMID 24991834
- [Background] Ghermezi M, Spektor TM, Berenson JR. The role of JAK inhibitors in multiple myeloma. Clin Adv Hematol Oncol. 2019 Sep;17(9):500-505. PMID 31549971
- [Background] de Oliveira MB, Fook-Alves VL, Eugenio AIP, Fernando RC, Sanson LFG, de Carvalho MF, Braga WMT, Davies FE, Colleoni GWB. Anti-myeloma effects of ruxolitinib combined with bortezomib and lenalidomide: A rationale for JAK/STAT pathway inhibition in myeloma patients. Cancer Lett. 2017 Sep 10;403:206-215. doi: 10.1016/j.canlet.2017.06.016. Epub 2017 Jun 20. PMID 28645562
- [Background] Tian Z, D'Arcy P, Wang X, Ray A, Tai YT, Hu Y, Carrasco RD, Richardson P, Linder S, Chauhan D, Anderson KC. A novel small molecule inhibitor of deubiquitylating enzyme USP14 and UCHL5 induces apoptosis in multiple myeloma and overcomes bortezomib resistance. Blood. 2014 Jan 30;123(5):706-16. doi: 10.1182/blood-2013-05-500033. Epub 2013 Dec 6. PMID 24319254
- [Background] Das DS, Das A, Ray A, Song Y, Samur MK, Munshi NC, Chauhan D, Anderson KC. Blockade of Deubiquitylating Enzyme USP1 Inhibits DNA Repair and Triggers Apoptosis in Multiple Myeloma Cells. Clin Cancer Res. 2017 Aug 1;23(15):4280-4289. doi: 10.1158/1078-0432.CCR-16-2692. Epub 2017 Mar 7. PMID 28270494
- [Background] Song Y, Li S, Ray A, Das DS, Qi J, Samur MK, Tai YT, Munshi N, Carrasco RD, Chauhan D, Anderson KC. Blockade of deubiquitylating enzyme Rpn11 triggers apoptosis in multiple myeloma cells and overcomes bortezomib resistance. Oncogene. 2017 Oct 5;36(40):5631-5638. doi: 10.1038/onc.2017.172. Epub 2017 Jun 5. PMID 28581522
- [Background] Peterson LF, Sun H, Liu Y, Potu H, Kandarpa M, Ermann M, Courtney SM, Young M, Showalter HD, Sun D, Jakubowiak A, Malek SN, Talpaz M, Donato NJ. Targeting deubiquitinase activity with a novel small-molecule inhibitor as therapy for B-cell malignancies. Blood. 2015 Jun 4;125(23):3588-97. doi: 10.1182/blood-2014-10-605584. Epub 2015 Mar 26. PMID 25814533
- [Background] Wang X, Mazurkiewicz M, Hillert EK, Olofsson MH, Pierrou S, Hillertz P, Gullbo J, Selvaraju K, Paulus A, Akhtar S, Bossler F, Khan AC, Linder S, D'Arcy P. The proteasome deubiquitinase inhibitor VLX1570 shows selectivity for ubiquitin-specific protease-14 and induces apoptosis of multiple myeloma cells. Sci Rep. 2016 Jun 6;6:26979. doi: 10.1038/srep26979. PMID 27264969
- [Background] Driessen C, Muller R, Novak U, Cantoni N, Betticher D, Mach N, Rufer A, Mey U, Samaras P, Ribi K, Besse L, Besse A, Berset C, Rondeau S, Hawle H, Hitz F, Pabst T, Zander T. Promising activity of nelfinavir-bortezomib-dexamethasone in proteasome inhibitor-refractory multiple myeloma. Blood. 2018 Nov 8;132(19):2097-2100. doi: 10.1182/blood-2018-05-851170. Epub 2018 Sep 20. No abstract available. PMID 30237154
- [Background] Richardson PG, Wolf J, Jakubowiak A, Zonder J, Lonial S, Irwin D, Densmore J, Krishnan A, Raje N, Bar M, Martin T, Schlossman R, Ghobrial IM, Munshi N, Laubach J, Allerton J, Hideshima T, Colson K, Poradosu E, Gardner L, Sportelli P, Anderson KC. Perifosine plus bortezomib and dexamethasone in patients with relapsed/refractory multiple myeloma previously treated with bortezomib: results of a multicenter phase I/II trial. J Clin Oncol. 2011 Nov 10;29(32):4243-9. doi: 10.1200/JCO.2010.33.9788. Epub 2011 Oct 11. PMID 21990396
- [Background] Castaigne S, Lefebvre P, Chomienne C, Suc E, Rigal-Huguet F, Gardin C, Delmer A, Archimbaud E, Tilly H, Janvier M, et al. Effectiveness and pharmacokinetics of low-dose all-trans retinoic acid (25 mg/m2) in acute promyelocytic leukemia. Blood. 1993 Dec 15;82(12):3560-3. PMID 8260694
- [Background] Zhou H, Lee JJ, Yuan Y. BOP2: Bayesian optimal design for phase II clinical trials with simple and complex endpoints. Stat Med. 2017 Sep 20;36(21):3302-3314. doi: 10.1002/sim.7338. Epub 2017 Jun 7. PMID 28589563
- [Background] Perel G, Bliss J, Thomas CM. Carfilzomib (Kyprolis): A Novel Proteasome Inhibitor for Relapsed And/or Refractory Multiple Myeloma. P T. 2016 May;41(5):303-7. No abstract available. PMID 27162470
- See also: Bayesian Optimal Interval Designs for Phase I Clinical Trials — https://odin.mdacc.tmc.edu/~yyuan/Software/BOIN/paper.pdf
- See also: Continued Improvement in Survival of Patients with Newly Diagnosed Multiple Myeloma (MM) — https://ash.confex.com/ash/2020/webprogram/Paper140388.html